CLINICAL TRIAL: NCT01836211
Title: High-Sensitivity Troponin T and Coronary Computed Tomography Angiography for Rapid Diagnosis of Emergency Chest Pain: a Randomized Controlled Study
Brief Title: High-Sensitivity Troponin T and Coronary Computed Tomography Angiography for Rapid Diagnosis of Emergency Chest Pain
Acronym: TRUE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IIBSP-DIA-2010-18
Record Dates: First submitted 2012-11-23; First posted 2013-04-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Chest Pain; Acute Coronary Syndrome
Keywords: Chest pain; Acute coronary syndrome; Cardiac biomarkers; Computed coronary tomography angiography; Emergency department
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fast strategy (Experimental): High sensitivity cardiac troponin T followed by computed coronary tomography angiography
  Interventions: Other: Fast strategy
- Standard of care strategy (Active Comparator): Standard of care strategy based on serial electrocardiograms and cardiac biomarkers followed by stress/rest cardiac imaging study
  Interventions: Other: Standard of care strategy

INTERVENTIONS:
Other: Fast strategy — High sensitivity troponin T followed by computed coronary tomography angiography
  Arms: Fast strategy
Other: Standard of care strategy — Standard of care strategy: serial electrocardiograms and cardiac biomarkers followed by stress/rest cardiac imaging study
  Arms: Standard of care strategy

SUMMARY:
* The purpose of this study is to determine the efficacy and safety of an evaluation strategy based on utilization of high sensitivity cardiac troponin T (hscTnT), followed by coronary computed tomography angiography (CCTA) in patients with low-intermediate risk chest pain consistent with a possible acute coronary syndrome compared to a standard of care (SOC) strategy.
* Unicentric, randomized, controlled, open label clinical trial that will compare a fast strategy (hscTnT followed by CCTA) with a SOC strategy (serial ECG and cardiac biomarkers followed by stress/rest imaging study).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chest pain consistent with possible acute coronary syndrome.
* Age > 18 years.
* Informed consent.

Exclusion Criteria:

* Previous history of coronary artery disease.
* Electrocardiogram diagnostic or suggestive of myocardial ischemia.
* Condition other than coronary artery disease as cause of an imbalance between myocardial oxygen supply and/or demand (eg. anemia, fever, arrhythmias).
* Chronic kidney disease (GFR <30 mL/min/1,73 m2).
* Iodine contrast allergy.
* Incapability to perform treadmill stress test.
* Barthel activity of daily living scale index < 100.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
All cause mortality, new myocardial infarction, new unstable angina, new heart failure, new hospital admission, new consult to the Emergency Department | 1 month after index event
  Composite end-point.

SECONDARY OUTCOMES:
All cause mortality | 1 month
Myocardial infarction | 1 month
Unstable angina | 1 month
Heart Failure | 1 month
Hospital admission | 1 month
  New cardiovascular hospital admission

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Cruz y San Pablo, Barcelona, Barcelona, Spain